CLINICAL TRIAL: NCT00299260
Title: A Phase II Immunogenicity Trial of Cytomegalovirus Glycoprotein B Vaccine in Allograft Candidate Recipients
Brief Title: CMV Glycoprotein B Vaccine in Allograft Recipients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Prof Paul Griffiths, University College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 04-107; R01AI051355 (NIH)
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2008-01

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus, glycoprotein B vaccine, allograft
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vaccine (Active Comparator): glycoprotein B plus MF59 adjuvant
  Interventions: Biological: CMV gB vaccine
- placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CMV gB vaccine — 20 micrograms
  Arms: vaccine
Drug: Placebo — normal saline
  Arms: placebo

SUMMARY:
Patients who receive transplants are at increased risk of developing serious cytomegalovirus (CMV) infections because they have a decreased immune system. The purpose of this study is to evaluate the safety and immune response of a CMV vaccine in patients (18 years old and older) who are awaiting a transplant. Following immunization with vaccine or placebo (inactive substance), patients will be followed for the development of immune responses to CMV and for evidence of CMV infection following transplantation. One hundred forty eligible patients will receive 3 injections of the CMV gB vaccine or 3 doses of placebo during 5 visits. Participants will participate in the study for approximately 7 months (if they do not undergo a transplant) or 10 months (if they undergo a transplant).

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is a common infectious agent which is well adapted to survival in the normal human host. Although CMV infection is usually asymptomatic, CMV disease develops when the host: virus balance is perturbed. This may occur when individuals become immunocompromised as a result of immunosuppressive drugs required to maintain an allograft. Currently there is no vaccine for the prevention of CMV infection. To reduce the impact of CMV infection, allograft transplant patients are either given prophylaxis with antiviral drugs or preemptive anti CMV therapy is given as soon as there is some indication of a productive infection from serial samples of blood. The primary objectives of this study are: to determine if recombinant soluble glycoprotein B cytomegalovirus vaccine is immunogenic when administered to patients awaiting transplantation of a kidney or liver; and to describe the safety profile of a 0-, 1-, and 6-month schedule of the CMV gB vaccine in patients awaiting transplantation. The secondary observational objectives of this study are: to determine if prior receipt of vaccine can reduce the incidence or quantity or cytomegalovirus DNA detection in the blood post transplant among patients who proceed to transplantation; to determine if prior receipt of vaccine does reduce the incidence or quantity of CMV DNA detected in the blood post transplant, to determine if the titer of neutralizing antibody induced after completing the course of immunization is a correlate of this immune protection; to describe the persistence of vaccine-induced neutralizing antibody, including the time when patients are given immunosuppressive drugs required for transplantation; to determine if prior receipt of vaccine does reduce the incidence or quantity of CMV DNA detected in the blood post transplant, to determine if the titer of neutralizing antibody present at the time of transplant is a correlate of this immune protection; and to explore the CD8 and CD4 responses among patients who proceed to transplantation. This study is a phase II trial with a randomized, blind-observer, placebo-controlled design. Patients will receive 3 injections each of 20 micrograms of the CMV gB vaccine or 3 doses of placebo. Participants will include 140 eligible patients (70 seronegative, 70 seropositive). Randomization will be stratified into 4 groups as follows; approximately 42 seronegative renal patients; approximately 42 seropositive renal patients; approximately 28 seronegative liver patients; approximately 28 seropositive liver patients. Serious adverse events (SAEs) will be followed until 1 month after the last vaccination and suspected unexpected serious adverse reactions (SUSARs) at any time during the follow-up period until 90 days post-transplant. The primary immunogenicity endpoints include: level of antibody by ELISA anti-gB at Days 0, 28, 56, 180, and 208 [ELISA Anti-gB (IgG) and CMV neutralizing antibody titers which will be assessed at each of the following timepoints: before and one month after the first vaccination; before and one month after the second vaccination; and before and one month after the third vaccination.]; and titer of neutralizing antibody at Days 0, 28, 56, 180, and 208. The primary safety endpoint will be the occurrence, severity, onset, and duration of injection site reactions or systemic reactions/events within 28 days following each injection and SUSARs at any time during the follow-up period until 90 days post-transplant. The observational endpoints measured in patients who proceed to transplant will include: increase of viral load (AUC/d) among those who become PCR positive during the 90 day follow-up post transplant; titer of neutralizing antibody detected at the time of transplant and at Days 0, 7, 35, 63, and 90 post transplant; and CD8 and CD4 responses at Days 0, 7, 35, 63, and 90 post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and/or assent must be obtained from the patient.
* Patients must be 18 years of age or older.
* Awaiting a liver or kidney transplant.
* All female patients with childbearing potential must have a negative pregnancy test prior to each vaccination.
* All females of childbearing potential must agree to use an effective barrier method of birth control while receiving the vaccine and for 30 days after completion of the course of vaccine. Other contraception in addition to barrier methods is permitted.
* Among the CMV seropositives, HLA type compatible with tetramer assays (currently A2, A24, B7, B8, B35). (seronegatives of any HLA type are eligible).

Exclusion Criteria:

* Patient unable or unwilling to provide and sign an informed consent or assent.
* If a patient who is competent to give informed consent enters the trial but subsequently becomes incompetent, they will be withdrawn.
* Pregnant or breastfeeding females.
* Participation in another clinical trial of a vaccine or of a systemic drug in the 4 weeks preceding the first trial vaccination (participation in trials of medical devices/ procedures is allowed).
* Planned participation in another clinical trial of a vaccine or of a systemic drug during the present trial period (participation in trials of medical devices/ procedures is allowed).
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Blood or blood-derived products received in the past 3 months (except albumin).
* Current thrombocytopenia or bleeding disorder contraindicating IM vaccination.
* Among the seropositives, HLA type incompatible with tetramer assays (seronegatives of any HLA type are eligible).
* Requiring emergency transplant for fulminant liver failure.
* Patients known to be HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
safety | 28 days
  SAEs within 28 days of each vaccine dose
immunogenicity | day 56
  antibody level one month after second dose of vaccine

SECONDARY OUTCOMES:
viral load | 90 days
  viral load in first 90 days post transplant
correlate of immune protection | 90 days
  correlation between antibody levels and viral load

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Griffiths, MD DSc, Principal Investigator — University College, London
Locations (1):
- University College Medical School, London, United Kingdom

REFERENCES:
- [Derived] Griffiths PD, Stanton A, McCarrell E, Smith C, Osman M, Harber M, Davenport A, Jones G, Wheeler DC, O'Beirne J, Thorburn D, Patch D, Atkinson CE, Pichon S, Sweny P, Lanzman M, Woodford E, Rothwell E, Old N, Kinyanjui R, Haque T, Atabani S, Luck S, Prideaux S, Milne RS, Emery VC, Burroughs AK. Cytomegalovirus glycoprotein-B vaccine with MF59 adjuvant in transplant recipients: a phase 2 randomised placebo-controlled trial. Lancet. 2011 Apr 9;377(9773):1256-63. doi: 10.1016/S0140-6736(11)60136-0. PMID 21481708